CLINICAL TRIAL: NCT01566617
Title: Impact of The Pharmaceutical Care on the Quality of Life of Patients With Chagas Disease and Heart Failure: Randomized Clinical Trial
Brief Title: Impact of the Pharmaceutical Care on the Quality of Life in Patients With Chagas Heart Disease
Acronym: ChagasCare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evandro Chagas Institute of Clinical Research (Other)
Collaborators: Alejandro Marcel Hasslocher Moreno, MD MSc PhD student (Unknown); Andrea Costa, MD PhD (Unknown); Andrea Silvestre de Sousa, MD PhD (Unknown); Luiz Henrique C. Sangenis, MD MSc PhD student (Unknown); Marcelo Teixeira de Holanda, MD MSc PhD student (Unknown); Mayara da Costa Chambela - MSc student (Unknown); Pedro Emmanuel Alvarenga Americano do Brasil, MD PhD (Unknown); Roberto Magalhães Saraiva, MD PhD (Unknown); Sergio Salles Xavier, MD PhD (Unknown)
Responsible Party: Principal Investigator, Gilberto Marcelo Sperandio da Silva, PhD, Evandro Chagas Institute of Clinical Research
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Chagas2303; 0034.0.009.000-11 (Other: Research Ethics Committee of the Evandro Chagas Clinical Research Institute (IPEC))
Record Dates: First submitted 2012-03-23; First posted 2012-03-29 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Chagas Heart Disease
MeSH Terms: interventions — Standard of Care; Pharmaceutical Services

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Other): (1) group who will receive standard care
  Interventions: Other: Standard care
- Standard Care and Pharmaceutical Care (Other): (2) group who will receive standard care and pharmaceutical care
  Interventions: Other: Standard care and Pharmaceutical care

INTERVENTIONS:
Other: Standard care and Pharmaceutical care — Pharmaceutical care is the direct interaction between the pharmacist and the drug's users in order to improve the therapeutic compliance among outpatients and promote adequate pharmacotherapeutic follow-up.
  Arms: Standard Care and Pharmaceutical Care
Other: Standard care — These patients will only receive standard care, with out follow-up by the pharmacist
  Arms: Standard Care

SUMMARY:
The investigators hypothesize that pharmaceutical care may constitute an important tool for the clinical management of these patients by improving their compliance to their treatment with consequent improvement in their quality of life by minimizing symptoms, and decreasing the number of hospital admissions and adverse drug reactions. Therefore, the aim of this trial is to evaluate the contribution of pharmaceutical care to clinical treatment of patients with Chagas heart disease complicated by heart failure.

Study Type: Interventional

Study Design: A total of 88 patients will be randomly assigned into two parallel groups: (1) group who will receive standard care and pharmaceutical care; and (2) group who will receive only standard care. Both groups will be subjected to a follow-up period of 12 months. The primary outcome of this trial is the evaluation of quality of life, measured by the 36-item short-form and the Minnesota Living with Heart Failure Questionnaire. Secondary outcomes include drug-related problems and exercise tolerance measured by the standard six-minute walk test.

ELIGIBILITY:
Inclusion Criteria:

* The proposed clinical trial will be conducted in volunteers with Chagas disease complicated by heart failure.
* Subjects will include adults, men and women, racial or ethnic minorities.
* Diagnosed by two distinct Chagas serology tests (indirect immunofluorescence and enzyme linked immunosorbent assay

Exclusion Criteria:

* Patients with any of comorbidities that significantly affect the cardiac performance, such as coronary artery disease, moderate or severe heart valvular disease, left ventricular (LV) hypertrophy, congenital heart disease, or that limit their survival, such as malignant tumors and HIV, will be excluded from the study.
* Patients will be also be excluded in case of failure to give informed consent, inability to perform 6 minute- walk test, significant cognitive impairment, or pregnancy.
* Individuals who are participating in others intervention trials will also be excluded.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Quality of life. | 12 months
  The primary outcome of this trial is the evaluation of quality of life, measured by the 36-item short-form and the Minnesota Living with Heart Failure Questionnaire. Evaluation of patient quality of life during follow up of two parallel groups: (1) group who will receive standard care and pharmaceutical care; and (2) group who will receive only standard care.

SECONDARY OUTCOMES:
Incidence and types of drug-related problems | 12 months
  To evaluate the drug-related problems based on the classiﬁcation of the Brazilian Pharmaceutical Care Consensus. Evaluation of drug-related problems during follow up of two parallel groups: (1) group who will receive standard care and pharmaceutical care; and (2) group who will receive only standard care.
Physical functional capacity. | 12 months
  All patients will have their physical functional capacity measured by the 6 minute-walk test (The patients will split in two parallel groups: (1) group who will receive standard care and pharmaceutical care; and (2) group who will receive only standard care). The test will be performed at the beginning of protocol and after 12 months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto M Silva, pharmaceutical, Principal Investigator — Evandro Chagas Clinical Research Institute
Locations (1):
- Evandro Chagas Clinical Research Institute, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Sperandio da Silva GM, Chambela MC, Sousa AS, Sangenis LH, Xavier SS, Costa AR, Brasil PE, Hasslocher-Moreno AM, Saraiva RM. Impact of pharmaceutical care on the quality of life of patients with Chagas disease and heart failure: randomized clinical trial. Trials. 2012 Dec 27;13:244. doi: 10.1186/1745-6215-13-244. PMID 23270509